CLINICAL TRIAL: NCT04690413
Title: NOWDx Test for the Detection of Antibodies to COVID-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NOWDiagnostics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NOWDx COVID-19 Antibody POC
Record Dates: First submitted 2020-08-31; First posted 2020-12-30 (Actual); Results first posted 2022-10-28 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2022-10

CONDITIONS: COVID-19; SARS-CoV-2; Coronavirus
MeSH Terms: conditions — COVID-19; Coronavirus Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Persons tested with investigational device (Experimental): Persons tested with investigational device who previously tested positive or negative for COVID-19 with an emergency use authorized or FDA cleared COVID-19 test
  Interventions: Device: NOWDx COVID-19 Test

INTERVENTIONS:
Device: NOWDx COVID-19 Test — The investigational device is the NOWDx COVID-19 Test.

SUMMARY:
This study is designed to compare the performance of the NOWDx COVID-19 Test to an emergency use authorized PCR test result. The intent is to show the rapid test device is comparable to a currently marketed device. The NOWDx COVID-19 Test is an in vitro lateral flow immunoassay intended for qualitative detection of total antibodies to SARS-CoV-2 in human whole blood (venous and fingerstick).

DETAILED DESCRIPTION:
This study is designed to compare the performance of the NOWDx COVID-19 Test to an emergency use authorized PCR test result. The intent is to show the rapid test device is comparable to a currently marketed device. The NOWDx COVID-19 Test is an in vitro lateral flow immunoassay intended for qualitative detection of total antibodies to SARS-CoV-2 in human whole blood (venous and fingerstick).

The NOWDx COVID-19 Test is intended for use as an aid in identifying individuals with an adaptive immune response to SARS-CoV-2, indicating recent or prior infection. At this time, it is unknown for how long antibodies persist following infection and if the presence of antibodies confers protective immunity. Testing of human venous whole blood (EDTA) and fingerstick specimens are intended to be conducted in patient care settings authorized to perform CLIA waived tests.

ELIGIBILITY:
Inclusion Criteria:

* Persons ≥18 years old;
* Persons who have tested positive or negative (within 6 days) for COVID-19 with an emergency use authorized molecular (PCR) test and can furnish said test report.

Exclusion Criteria:

* Persons <18 years old;
* Persons who have previously participated in a NOWDx study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Beth L Cobb, Principal Investigator — NOWDiagnostics, Inc.
Locations (3):
- United States (3):
  - Del Sol Research Management, LLC, Tucson, Arizona
  - Comprehensive Clinical Research, LLC, West Palm Beach, Florida
  - Clinical Research Solutions, LLC, Jackson, Tennessee

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Persons Tested With Investigational Device
Started | 129
Completed | 124
Not Completed | 5

BASELINE CHARACTERISTICS:
Arm/Group | Persons Tested With Investigational Device
Number analyzed (Participants) | 124
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 114
  >=65 years | 10
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 74
  Male | 50
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 30
  Not Hispanic or Latino | 88
  Unknown or Not Reported | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 52
  White | 64
  More than one race | 2
  Unknown or Not Reported | 5
Region of Enrollment [Number; unit: participants]
  United States | 124

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Clinical Agreement Between NOWDx COVID-19 Test and Emergency Use Authorized or FDA Cleared Comparator.
Description: Calculate positive percent agreement (PPA) and negative percent agreement (NPA) between NOWDx COVID-19 Test and emergency use authorized or FDA cleared COVID-19 PCR Test.
Time Frame: 1 day
Measure: Number; unit: percentage of results matching PCR
Arm/Group | Persons Tested With Investigational Device
Number analyzed (Participants) | 124
percentage of results matching PCR
  PPA | 91.5
  NPA | 95.4

ADVERSE EVENTS:
Time Frame: Sites were required to report adverse events to the Sponsor within 10 days. Serious adverse events were required to be reported to the Sponsor within 24 hours. All adverse event data were required to be collected through study completion, an average of 4 months.
Arm/Group | Persons Tested With Investigational Device
All-Cause Mortality (participants affected / at risk) | 0/124
Serious Adverse Events (participants affected / at risk) | 0/124
Other Adverse Events (participants affected / at risk) | 0/124

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-07-22): https://cdn.clinicaltrials.gov/large-docs/13/NCT04690413/Prot_000.pdf
  • Statistical Analysis Plan (2020-09-01): https://cdn.clinicaltrials.gov/large-docs/13/NCT04690413/SAP_001.pdf